CLINICAL TRIAL: NCT06238947
Title: LONG-TERM EVALUATION OF OUTCOMES OF PATIENTS UNDERGOING AUTOLOGOUS CHONDROCYTE TRANSPLANTATION DELIVERED ON BIOMATERIAL (HYALOGRAFT C) Prospective Observational Study
Brief Title: Long-term Outcome Evaluation of Patients Undergoing Autologous Chondrocyte Transplantation Delivered on Biomaterial
Status: Not yet recruiting | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: Chondro-Long
Record Dates: First submitted 2024-01-26; First posted 2024-02-02 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Cartilage Injury; Cartilage Disease
Keywords: autologous chondrocyte transplantation; osteochondral defects
MeSH Terms: conditions — Cartilage Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Chondro-Long study is prospective observational study for a long-term clinical evaluation (follow-up up to 25 years) in patients treated with autologous chondrocyte transplantation delivered on biomaterial for full-thickness chondral defects (Outerbridge grade III - IV) at the level of femoral condyles, trochlea, patella and tibial plateau.

The aim of the study is to collect long-term clinical data from the case series of patients surgically treated from 1999 to 2006 with autologous chondrocyte transplantation delivered on biomaterial for full-thickness chondral defects (Outerbridge grade III - IV) or osteochondral defects at the level of femoral condyles, trochlea, patella, and tibial plateau. The objective of the study is to demonstrate the efficacy of this long-term cartilage regeneration technique (follow-up up to 25 years) in improving patient symptomatology and functional capacity

DETAILED DESCRIPTION:
Patients will be recruited from all subjects surgically treated with autologous chondrocyte transplantation delivered on biomaterial for chondral/osteochondral lesions at the femoral condyles, trochlea, patella, and tibial plateau from 1999 to 2006 at the Rizzoli Orthopaedic Institute. The study has 3 phases: Identification of includable patients, Follow-up assessment byTelemedicine platform, and the collection of study-specific clinical data of enrolled patients.

Clinical score data will be collected from the medical records and questionnaires conducted in the mid-term of patients enrolled in the study. These data will be used, together with data collected by telemedicine/long-term e-mail questionnaire, to evaluate the time course of outcomes after surgical treatment with autologous chondrocyte transplantation delivered on biomaterial

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent autologous chondrocyte transplantation surgery delivered on biomaterial (Hyalograft C) from 1999 to 2006 at the Rizzoli Orthopaedic Institute who met the following criteria at the time of surgery:
* Full-thickness chondral defects (Outerbridge grade III - IV) and osteochondral defects at the femoral condyles, trochlea, patella and tibial plateau.
* Patients aged between 14 and 60 years at the time of surgery.
* Male and female sex.

Exclusion Criteria:

* Patients no longer available

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients treated with autologous chondrocyte transplantation delivered on biomaterial (Hyalograft C, Fidia, Abano Terme ) for full-thickness chondral defects (Outerbridge grade III to IV) at the level of femoral condyles, trochlea, patella, and tibial plateau
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score (IKDC)-Subjective Knee Evaluation Form | baseline
  This is a subjective, knee-specific rating scale that is considered one of the most reliable assessment tools in the evaluation of knee pathology. The questionnaire examines 3 categories: symptoms, sports activity, and knee function. According to this questionnaire, a score between 0 and 100 can be obtained, where a high score is associated with a high level of function and minor pain symptoms. A score of 100 is in fact interpreted as a condition in which there are neither limitations in conducting activities of daily living nor symptoms
EuroQol Visual Analogue Scale (EQ-VAS ) | baseline
  This is a visual analog scale that has a range of scores from 0 (worst imaginable health condition) to 100 (best imaginable health condition).
Tegner Score | baseline
  This questionnaire allows the estimation of a subject's motor activity level with a score between 0 and 10, where 0 represents 'inability' and 10 represents 'participation in competitive sports, such as soccer at the national or international level. This score is the one most commonly used to define the motor activity level of patients with knee disorders. In the study, the Tegner Score will be filled in directly by the investigator, through an interview the patient. In addition, questions will also be asked about return to sports and pre-injury, pre-treatment and recovered/achieved sports level .
EQ-5D (EuroQoL) Current Health Assessment | baseline
  EQ-5D is a standardized measure of health-related quality of life developed by the EuroQol Group to provide a simple generic questionnaire for use in clinical and economic evaluation and population health surveys
MCD/MCID (Minimal Clinically Important Difference): | baseline
  the patient should indicate satisfaction and relative degree of improvement for the treatment performed
Patient Acceptable Symptom State (PASS) | baseline
  A tool to assess patient satisfaction in consideration of their current degree of pain, function, and daily activity. Patients can express if their state of health will be satisfying, answering "yes" or "no.

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Zaffagnini, MD, Principal Investigator — Istituto Ortopedico Rizzoli - II Clinica Ortopedica e Traumatologica

REFERENCES:
- [Background] Anderson AF, Irrgang JJ, Kocher MS, Mann BJ, Harrast JJ; International Knee Documentation Committee. The International Knee Documentation Committee Subjective Knee Evaluation Form: normative data. Am J Sports Med. 2006 Jan;34(1):128-35. doi: 10.1177/0363546505280214. Epub 2005 Oct 11. PMID 16219941
- [Background] Aroen A, Loken S, Heir S, Alvik E, Ekeland A, Granlund OG, Engebretsen L. Articular cartilage lesions in 993 consecutive knee arthroscopies. Am J Sports Med. 2004 Jan-Feb;32(1):211-5. doi: 10.1177/0363546503259345. PMID 14754746
- [Background] Bauer S, Khan RJ, Ebert JR, Robertson WB, Breidahl W, Ackland TR, Wood DJ. Knee joint preservation with combined neutralising high tibial osteotomy (HTO) and Matrix-induced Autologous Chondrocyte Implantation (MACI) in younger patients with medial knee osteoarthritis: a case series with prospective clinical and MRI follow-up over 5 years. Knee. 2012 Aug;19(4):431-9. doi: 10.1016/j.knee.2011.06.005. Epub 2011 Jul 22. PMID 21782452
- [Background] Behrens P, Bitter T, Kurz B, Russlies M. Matrix-associated autologous chondrocyte transplantation/implantation (MACT/MACI)--5-year follow-up. Knee. 2006 Jun;13(3):194-202. doi: 10.1016/j.knee.2006.02.012. Epub 2006 Apr 24. PMID 16632362
- [Background] Della Villa S, Kon E, Filardo G, Ricci M, Vincentelli F, Delcogliano M, Marcacci M. Does intensive rehabilitation permit early return to sport without compromising the clinical outcome after arthroscopic autologous chondrocyte implantation in highly competitive athletes? Am J Sports Med. 2010 Jan;38(1):68-77. doi: 10.1177/0363546509348490. PMID 20051508
- [Background] de Windt TS, Bekkers JE, Creemers LB, Dhert WJ, Saris DB. Patient profiling in cartilage regeneration: prognostic factors determining success of treatment for cartilage defects. Am J Sports Med. 2009 Nov;37 Suppl 1:58S-62S. doi: 10.1177/0363546509349765. PMID 19934438
- [Background] Ebert JR, Robertson WB, Woodhouse J, Fallon M, Zheng MH, Ackland T, Wood DJ. Clinical and magnetic resonance imaging-based outcomes to 5 years after matrix-induced autologous chondrocyte implantation to address articular cartilage defects in the knee. Am J Sports Med. 2011 Apr;39(4):753-63. doi: 10.1177/0363546510390476. Epub 2011 Jan 21. PMID 21257846
- [Background] Ferruzzi A, Buda R, Faldini C, Vannini F, Di Caprio F, Luciani D, Giannini S. Autologous chondrocyte implantation in the knee joint: open compared with arthroscopic technique. Comparison at a minimum follow-up of five years. J Bone Joint Surg Am. 2008 Nov;90 Suppl 4:90-101. doi: 10.2106/JBJS.H.00633. No abstract available. PMID 18984722
- [Background] Filardo G, Kon E, Andriolo L, Vannini F, Buda R, Ferruzzi A, Giannini S, Marcacci M. Does patient sex influence cartilage surgery outcome? Analysis of results at 5-year follow-up in a large cohort of patients treated with Matrix-assisted autologous chondrocyte transplantation. Am J Sports Med. 2013 Aug;41(8):1827-34. doi: 10.1177/0363546513480780. Epub 2013 Jul 15. PMID 23857885
- [Background] Andriolo L, Reale D, Di Martino A, De Filippis R, Sessa A, Zaffagnini S, Filardo G. Long-term Results of Arthroscopic Matrix-Assisted Autologous Chondrocyte Transplantation: A Prospective Follow-up at 15 Years. Am J Sports Med. 2020 Oct;48(12):2994-3001. doi: 10.1177/0363546520949849. Epub 2020 Sep 16. PMID 32936677